CLINICAL TRIAL: NCT03476226
Title: Cognitive Dysfunction and the Breast Cancer Patient: A Study to Determine the Impact of Providing Information on Coping Strategies on Quality of Life
Brief Title: Cognitive Dysfunction and Breast Cancer Coping Strategies Impact on QOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6727
Record Dates: First submitted 2018-03-01; First posted 2018-03-26 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Quality of Life; Cognitive Dysfunction; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The research team will provide the intervention to subjects. Intervention: The nursing-driven Cognitive Dysfunction Coping Strategy Teaching Sheet and provide education as to its use.
  QOL survey administered
  Interventions: Other: Cognitive Dysfunction Coping Strategy Teaching Sheet
- Group 2 (No Intervention): Provide current standard of education for cognitive dysfunction. QOL survey administered

INTERVENTIONS:
Other: Cognitive Dysfunction Coping Strategy Teaching Sheet — Demographic sheet, Fact-Cog3, and teaching tool at baseline then week 4 and 8 Fact Cog3 and reinforcement of tool, at week 16 evaluation and Fact-Cog3
  Arms: Group 1

SUMMARY:
The purpose of this study is to determine whether patients experience a better quality of life when they have received education about coping strategies for cognitive dysfunction.

DETAILED DESCRIPTION:
Cancer treatment may consist of chemotherapy, radiation, hormone therapy, surgery or a combination of all disciplines. However, breast cancer therapies have at times demonstrated distressing effects in patients/survivors during and/or following treatment. One area that is found to cause distress for the breast cancer patient is changes in cognitive function.

Areas most commonly impacted by changes in cognitive function as a result of chemotherapy include executive functioning (including judgment, hindsight and foresight), processing speed or reaction time, working memory, and organizational skills.

Due to the limited amount of research involving quality of life as related to cognitive dysfunction, there is a clear need for additional investigation. Treatment typically focuses on the physical and psychosocial aspects of patients/survivors, however emphasis should also be placed on the impact of quality of life during treatment and survivorship due to the potential for far-reaching effects as previously discussed.

Oncology nurses may be instrumental in identifying patients with Cognitive Dysfunction. In doing so, the nurse may then communicate with the patient/survivor as to the impact of Cognitive Dysfunction on quality of life. The nurse can provide appropriate education and or additional support options.

ELIGIBILITY:
Inclusion Criteria:

* Age >18years old
* Stage 0-IV breast cancer (excluding stage IV with metastasis to the brain)
* Life expectancy > 3 months
* Able to speak and read English fluently
* Self-reported cognitive difficulties that interfere with everyday activities
* Reported Memory/Cognitive changes on Distress Thermometer
* Able to provide written and informed consent
* Willing to complete FACT-Cog questionnaire

Exclusion Criteria:

* Current Cognitive Training, for example, use of brain training, physical therapy, occupational or speech therapy for the sole purpose of improving cognitive function
* Recent diagnosis of Major depression or other current psychiatric disorders and are not considered stable per a current care provider
* History of Dementia or Alzheimer's Disease
* History of Central Nervous System (CNS) radiation, intrathecal chemotherapy, or CNS involved surgery
* History of metastatic disease extending to the brain
* History of traumatic brain injury
* History of seizure disorder
* History of thyroid disorder (Subjects that are well managed without changes in thyroid medications or doses for at least 6 months may participate in study)
* Current use of illicit substances and or alcohol (including medical marijuana)
* Current sleep disturbance/disorder (Subjects that are well managed without changes in sleep medications or doses for at least 6 months may participate in study).
* Concurrent use of antidepressants for example, use of antidepressants for pain management or smoking cessation. (Subjects that are well managed without changes on antidepressant medications or doses for at least 6 months may participate in study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
FACT-Cog 3 questionnaire | 16 weeks
  Assess QOL with use of FACT-Cog 3 questionnaire. Then compare group 1 that was provided teaching on coping strategies to Group 2 that received current standard of care. Determine impact on quality of life between subject groups based on statistical difference in Quality of Life between Group 1 and Group 2.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine L Szubski, BSN RN OCN, Principal Investigator — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois

IPD SHARING:
Plan to Share IPD: No